CLINICAL TRIAL: NCT01436617
Title: Assessing the Value of a Dosage of Anti-cetuximab in the Therapeutic Management of Patients With Colon Cancer or Upper Aero-digestive Tract and Candidates for Treatment With Cetuximab
Acronym: IgES
Status: Completed | Type: Observational
Sponsor: Centre Francois Baclesse (Other)
Collaborators: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: IgES
Record Dates: First submitted 2011-09-14; First posted 2011-09-19 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Colon Cancer; Head and Neck Cancer; Allergic Reaction
Keywords: cancer; colon; Head and neck; cetuximab; anti-cetuximab dosage
MeSH Terms: conditions — Colonic Neoplasms; Head and Neck Neoplasms; Hypersensitivity; Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: blood sample — The IgE anti cetuximab test will then be conducted by an ELISA test

SUMMARY:
The main objective of this study is to validate the utility of IgE anti-cetuximab in the treatment strategy to identify patients at risk for a severe allergic reaction to cetuximab (grade 3 or 4 of the classification of NCI) and thus reduce the incidence of severe reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent,
* Patient aged over 18 years
* Patients with a WHO performance status ≤ 2,
* Colon cancer or upper aero-digestive tract cytologically or histologically proven
* Patients with an indication to the theoretical use of cetuximab for colon neoplasia or upper aero-digestive tract,
* Haematological and biochemical compatible with combination therapy with cetuximab.

Exclusion Criteria:

* Patients previously treated with cetuximab,
* A person deprived of liberty or under supervision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer or upper aero-digestive tract and candidates for treatment with cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Validate the utility of an IgE anti-cetuximab test in the treatment strategy | 3 years
  We hypothesize that a positive specific IgE assay predicts the occurrence of an allergic reaction during the first dose of cetuximab. Thus, in population areas where the prevalence of specific IgE positive plasma is higher, the use of alternative therapies in patients with a positive test would reduce the incidence of anaphylactic reactions to cetuximab.
  If the use of specific IgE anti-cetuximab in the treatment strategy is effective, there will be reduction in the incidence of anaphylaxis to cetuximab in the participating centers.

CONTACTS AND LOCATIONS:
Overall Officials: GERVAIS Radj, MD, Principal Investigator — Centre François Baclesse
Locations (10):
- France (10):
  - CHU, Amiens
  - Centre hospitalier, Bayeux
  - CHU, Caen
  - Centre François Baclesse, Caen
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
  - CHU Charles Nicolle, Rouen
  - Centre Henri Becquerel, Rouen
  - Centre Paul Strauss, Strasbourg